CLINICAL TRIAL: NCT05730621
Title: A Study to Compare the Effects of Sarpogrelate Sustained Release /Aspirin Combination Therapy Versus Aspirin on Blood Viscosity in the Patients With Peripheral Arterial Disease and Coronary Artery Disease; A Prospective, Randomized, Parallel, Open-Label, Single-center, Phase IV Clinical Trial
Brief Title: A Study to Compare the Effects of Sarpogrelate Sustained Release /Aspirin Combination Therapy Versus Aspirin on Blood Viscosity in the Patients With Peripheral Arterial Disease and Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC047
Record Dates: First submitted 2023-01-26; First posted 2023-02-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Sarpogrelate; Blood Viscosity; Peripheral Arterial Disease; Coronary Artery Disease
Keywords: Sarpogrelate Sustained Release
MeSH Terms: conditions — Peripheral Arterial Disease; Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarpogrelate Sustained Release/Aspirin (Experimental): Sarpogrelate Sustained Release/Aspirin Combination Therapy for 12 weeks
  Interventions: Drug: Sarpogrelate Sustained Release/Aspirin
- Aspirin (Active Comparator): Aspirin Monotherapy qd for 12 weeks
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Sarpogrelate Sustained Release/Aspirin — Aspirin 100mg qd and Sarpogrelate Sustained Release 300mg qd for 12 weeks
  Arms: Sarpogrelate Sustained Release/Aspirin
Drug: Aspirin — Aspirin 100mg qd for 12 weeks
  Arms: Aspirin

SUMMARY:
This study is to compare the effects of sarpogrelate sustained release /aspirin combination therapy versus aspirin on blood viscosity in the patients with peripheral arterial disease and coronary artery disease

ELIGIBILITY:
Inclusion Criteria:

1. Both man and woman who is over 19 years old
2. Identified as 10-75% of Stenosis in Coronary Angiography or Coronary CTA(Coronary computed tomography angiography)
3. Patients who diagnosed with peripheral artery disease or has symptoms
4. Written informed consent

Exclusion Criteria:

1. Patients who is scheduled surgery due to coronary artery disease or cerebral infarction disease.
2. Patients who have taken aspirin within two weeks before randomization
3. Patients who need antiplatelet or anticoagulant medication except Aspirin
4. Confirmed below results at screening

   * Hemoglobin <13g/dL
   * Platelet <60,000/µL
   * Severe kidney disease patient with eGFR(estimated Glomerular Filtration Rate) <30 mL/min/1.73 m2 (CKD-EPI)
5. Patients with a history of cerebrovascular and cardiovascular complications (brain infarction, transient cerebral ischemic seizures, myocardial infarction, unstable angina, coronary artery bypass graft, percutaneous coronary artery intervention) within the last six months
6. Patients with bleeding
7. Pregnant or lactating women
8. Those participating in other clinical trials for investigational products
9. Patients deemed to be ineligible to participate in the trial by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 12 in Blood Viscosity(cP, centipoise) measured by the blood viscometer | Baseline/Week 12

SECONDARY OUTCOMES:
Change from baseline to week 4 in Blood Viscosity(cP, centipoise) measured by the blood viscometer | Baseline/Week 4
Change from baseline to week 4, 12 in Erythrocyte Deformability(elogation index at 3Pa) measured by Microfluidic Scanning Method | Baseline/Week 4/Week 12
Change from baseline to week 4, 12 in Erythrocyte Aggregation(critical shear stress) measured by Microfluidic Scanning Method | Baseline/Week 4/Week 12
Change from baseline to week 4, 12 in FMD(Flow Mediated Dilation) by Endothelium-dependent vasodilation measurement | Baseline/Week 4/Week 12
Rate of change from baseline to week 4, 12 in tODI(tissue oxygen delivery index) | Baseline/Week 4/Week 12
Proportion of subjects who tODI(tissue oxygen delivery index) have improved by 20% or more | Week 12
Rate of change from baseline to week 4, 12 in Lipid profile | Baseline/Week 4/Week 12
Rate of change from baseline to week 4, 12 in FPG(Fasting Plasma Glucose) | Baseline/Week 4/Week 12
Rate of change from baseline to week 4, 12 in HOMA-IR(Homeostatic Model Assessment for Insulin Resistance) | Baseline/Week 4/Week 12
Rate of change from baseline to week 4, 12 in hs-CRP(high sensitivity C-Reactive Protein) | Baseline/Week 4/Week 12
Change from baseline to week 12 in SF-36(Questionnaire for Medical Outcome Short Form Health Survey, 36-Item) | Baseline/Week 12
Change from baseline to week 12 in VAS(Visual Analogue Scale) | Baseline/Week 12

CONTACTS AND LOCATIONS:
Overall Officials: KeunSang Yum, Principal Investigator — The Catholic University of Korea Uijeongbu St. Mary's Hospital
Locations (1):
- The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No